CLINICAL TRIAL: NCT05415449
Title: Exploration of Central Venous Catheter Protective Devices in the Pediatric Population: A Mixed Methods Study
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Gus Gear Inc (Unknown); Society of Pediatric Nurses (Unknown)
Responsible Party: Principal Investigator, Maria Leal, Director of Acute Care Services, Children's Medical Center Dallas
Other Study IDs: STU-2022-0306
Record Dates: First submitted 2022-05-31; First posted 2022-06-13 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Central Line

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- No groups: Identify eligible patients--Informed Consent--Provide education and two protective wearable device--Demographic data (electronic health record)--Interview parent on device--Every month complete 30-day satisfaction survey for a total of three data collection period-Discharge from study.
  Nurse data collection scheme: Study participants hospitalized at time of enrollment in study or anytime during the study period. Nurse of patients using device will complete satisfaction survey.
  Interventions: Device: Gus gear protective wearable device

INTERVENTIONS:
Device: Gus gear protective wearable device — Gus gear protective wearable device for central line.

SUMMARY:
1. to determine the feasibility of utilizing a wearable device
2. to prospectively measure and evaluate parent and nurse satisfaction with the protective wearable device.

This is a sequential, convergent mixed methods study design in which qualitative interview data will be collected first followed by quantitative data.

Scheme and Outcomes: Identify eligible patients--Informed Consent--Provide education and two protective wearable device--Demographic data (electronic health record)--Interview parent on device--Every month complete 30-day satisfaction survey for a total of three data collection period-Discharge from study.

Nurse data collection scheme: Study participants hospitalized at time of enrollment in study or anytime during the study period. Nurse of patients using device will complete satisfaction survey.

Note: Vest is a Class I Exempt FDA-registered device.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CVCs ages 0 to 12 years of age
* May currently utilizing or historically utilized the interventional wearable protective device
* Caregiver or parent available
* English and Spanish speaking subjects

Exclusion Criteria:

* • Females with Tanner 2 breast or greater breast development. Justification: the wearable device will not fit properly to secure the CVC and may increase the risk of complications. If the patient does develop breast during the time of the study, then the patient will no longer wear the wrap and will go back to securing their device in the traditional way. Tanner 2 breast development will be evaluated in the screening process of patients.

  * Patients in critical care services such as neonates, trauma/ neurology intensive care unit, or cardiac intensive care unit. Justification: These patients are not mobile with their CVC and not the targeted population.

Ages: 0 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with CVCs ages 0 to 12 years of age
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Leal, BSN, RN, CPN, Principal Investigator — Children's Health UTSW
Locations (1):
- Children's Health, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- No Groups: As per protocol, there were 30 participants who were enrolled (they were all eligible and consented to the study). During the course of data collection, 6 out of 30 were unenrolled due to failed for follow-up/did not complete the data collection process.
  Identify eligible patients--Informed Consent--Provide education and two protective wearable device--Demographic data (electronic health record)--Interview parent on device--Every month complete 30-day satisfaction survey for a total of three data collection period-Discharge from study.
  Nurse data collection scheme: Study participants hospitalized at time of enrollment in study or anytime during the study period. Nurse of patients using device will complete satisfaction survey.
  Gus gear protective wearable device: Gus gear protective wearable device for central line.
Period: Overall Study
Arm/Group | No Groups
Started | 30
Completed | 24
Not Completed | 6
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- No Groups: Identify eligible patients--Informed Consent--Provide education and two protective wearable device--Demographic data (electronic health record)--Interview parent on device--Every month complete 30-day satisfaction survey for a total of three data collection period-Discharge from study.
  Nurse data collection scheme: Study participants hospitalized at time of enrollment in study or anytime during the study period. Nurse of patients using device will complete satisfaction survey.
  Gus gear protective wearable device: Gus gear protective wearable device for central line.
Arm/Group | No Groups
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 6 out of 30 were unenrolled
  Participants
    number analyzed (Participants) | 24
    Female | 14
    Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Population: 6 out of 30 were unenrolled
  Participants
    United States: number analyzed (Participants) | 24
    United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Measurement From Parents of Children Using the Gus Gear Vest Device
Description: No. of participants who were interviewed i.e. parents (of children using Gus gear vest) on device. Semi-structured interview guide was used to collect interview from parents. Eligible parents were parents of children between 0-12 years of age using the vest, and Parents should be able to speak English/Spanish. Interviews being qualitative in nature, the criteria to assess feasibility from parents using the vest will be done using transcription and inductive content analysis to find codes and themes from the data provided by the parents during the interview.
Time Frame: Two weeks from recruitment, plus or minus seven days.
Population: 30 is the enrolled number for quantitative piece of the study. Being mixed methods in nature in design, this study also has qualitative part. Upon interviewing 12 parents, thematic saturation was achieved to conclude data collection for the qualitative part of the study.
Measure: Number; unit: Interviews
Units Other Than Participants: interviews
Arm/Group | No Groups
Number analyzed (Participants) | 12
Number analyzed (interviews) | 12
Interviews | 12

2. Primary Outcome: Satisfaction Survey From Parents of Children Using the Gus Gear Vest Device
Description: Every month complete 30-day satisfaction survey for a total of three data collection period
Time Frame: Every month for a total of three data collection periods up to 3 months. Team will have plus or minus seven-day timeframe around the 30-day window to collect the data.
Reporting Status: Not Posted

3. Primary Outcome: Satisfaction Survey From Nurses
Description: Satisfaction survey from nurses of Children using the Gus gear vest device
Time Frame: Anytime during the study period up to nine months.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 months
Arm/Group | No Groups
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT05415449/Prot_SAP_000.pdf